CLINICAL TRIAL: NCT02209051
Title: A Multicenter, Prospective, Randomized, Parallel-group, Standard of Care-controlled Clinical Trial to Evaluate the Use of AMNIOEXCEL® in the Management of Chronic Diabetic Foot Ulcers
Brief Title: Phase IV Study to Evaluate the Efficacy of AMNIOEXCEL in Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS2014.01.01
Record Dates: First submitted 2014-07-31; First posted 2014-08-05 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Diabetic Foot Ulcers
Keywords: Diabetic Foot Ulcers; AMNIOEXCEL; Wagner Grade 1 or 2 foot ulcers; Wound; Foot health; Ulcer; Foot Ulcer; Diabetic Foot; Foot Diseases; Skin Diseases; Leg Ulcer; Skin Ulcer; Diabetic Angiopathies; Vascular Diseases; Cardiovascular Diseases; Diabetes Complications; Diabetes Mellitus; Endocrine System Diseases; Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Foot; Wounds and Injuries; Ulcer; Foot Ulcer; Foot Diseases; Skin Diseases; Leg Ulcer; Skin Ulcer; Diabetic Angiopathies; Vascular Diseases; Cardiovascular Diseases; Diabetes Complications; Diabetes Mellitus; Endocrine System Diseases; Diabetic Neuropathies | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMNIOEXCEL (Active Comparator): Human Amniotic Membrane Allograft
  Interventions: Other: AMNIOEXCEL; Other: Standard of Care, Diabetic Foot Ulcers
- Standard of Care, Diabetic Foot Ulcers (Active Comparator): Advanced wound care dressings and offloading of wound.
  Interventions: Other: Standard of Care, Diabetic Foot Ulcers

INTERVENTIONS:
Other: AMNIOEXCEL — Application of AMNIOEXCEL every 1-2 weeks for a period of 6 weeks or until wound closure, whichever is sooner.
  Arms: AMNIOEXCEL
Other: Standard of Care, Diabetic Foot Ulcers — Advanced wound care dressings and offloading applied daily for a period of 8 weeks or until wound closure

SUMMARY:
The primary goal of the study is to demonstrate the increased rate of complete wound closure by AMNIOEXCEL® compared to routine care in patients with chronic diabetic foot ulcers

DETAILED DESCRIPTION:
Potential study candidates will be Screened for Inclusion and Exclusion criteria after providing informed consent. Candidates will have their wound cleansed and debrided (if necessary), photographed and measured. Blood will be drawn for laboratory analyses. Patients will return two weeks later for assessment.

Upon return, per the original protocol, patient would have been randomized at <20% closure; per Amendment 1, if the wound has closed <30% in area during the 2 week Screening Period and all other eligibility criteria are met, the patient will be randomized (1:1) to receive either AMNIOEXCEL® with Standard of Care (SOC) or SOC alone.

All patients enrolled in this study will receive SOC. For the purposes of this study, Standard of Care (SOC) includes debridement of necrotic/non-viable tissue, moist wound dressings, off-loading (where appropriate, DH Walker only) and infection surveillance and management. For those randomized to receive AMNIOEXCEL®, in addition to SOC, the tissue will be applied after the wound has been debrided and hemostasis achieved. The wound will then be dressed with a non-adherent dressing (e.g. Adaptic) and covered with a moisture retentive dressing.

The patient will return once weekly for wound care, photographs and ulcer measurement. At each visit, the wound will be assessed and AMNIOEXCEL® reapplied as appropriate, based upon physician judgment. All patients complete their participation at Week 6.

This is an open label study and no attempt will be made to blind subjects or Investigators to randomization allocation.

ELIGIBILITY:
Inclusion Criteria:

1. an ambulatory person at least 18 years of age at the time of informed consent.
2. type 1 or type 2 diabetes mellitus.
3. glycosylated hemoglobin (HbA1c) of ≤12%
4. at least one wound that is/has:

   * Wagner grade 1 or superficial 2 (without bone, tendon or joint exposure),
   * duration of at least 1 month,
   * no clinical signs of infection or osteomyelitis,
   * between 1cm2 and 25cm2 in area,
   * per original protocol, closed <20% in area during the Screening Period; per Amendment #1, closed <30% in area during Screening and
   * located on the foot, distal to malleoli.
5. adequate circulation to the affected extremity
6. serum creatinine of <3.0mg/dl.

Exclusion Criteria:

1. participated in another clinical trial within 30 days prior to consent,
2. Active Charcot deformity of the study foot (i.e. erythematous, warm, edematous and actively remodeling)
3. receiving radiation or chemotherapy of any kind,
4. known or suspected malignancy of current ulcer,
5. pregnant or breast feeding,
6. an active malignant disease,
7. receiving hemo- or peritoneal dialysis,
8. sickle cell anemia or Raynaud's syndrome,
9. diagnosis of autoimmune connective tissue disease,
10. received a biologic agent, growth factor, xenograft or skin equivalent in the 30 days prior to consent,
11. exposed bone, tendon or joint capsule in the study ulcer,
12. currently receiving antibiotics (for any reason), or
13. taking medications considered to be immune system modulators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete wound closure (i.e. complete skin re-epithelialization without drainage or dressing requirements) at 6 weeks after initiation of study treatment | 8 weeks

SECONDARY OUTCOMES:
Time to complete wound closure of the target ulcer | 8 weeks
Rate of wound closure | 8 Weeks
Incidence, severity and type of adverse events | 8 Weeks
  This outcome measure represents a composite of collected adverse event data.
Changes in Quality of Life assessment | 8 Weeks

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Associated Foot and Ankle Specialists, LLC, Phoenix, Arizona
  - Center for Clinical Research, Inc., Castro Valley, California
  - Pacific Wound Center, Stockton, California
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Barry University Clinical Research, North Miami Beach, Florida
  - Beth Israel Deaconess Hospital - Plymouth, Plymouth, Massachusetts
  - Duke University, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina

REFERENCES:
- [Derived] Snyder RJ, Shimozaki K, Tallis A, Kerzner M, Reyzelman A, Lintzeris D, Bell D, Rutan RL, Rosenblum B. A Prospective, Randomized, Multicenter, Controlled Evaluation of the Use of Dehydrated Amniotic Membrane Allograft Compared to Standard of Care for the Closure of Chronic Diabetic Foot Ulcer. Wounds. 2016 Mar;28(3):70-7. PMID 26978860